CLINICAL TRIAL: NCT07075666
Title: Early Detection of Prostate Cancer Among Men in the Middle Region of Syria
Brief Title: Early Detection of Prostate Cancer of Syrian Men
Status: Enrolling by invitation | Type: Observational
Sponsor: Al-Hawash Private University (Other)
Responsible Party: Sponsor
Other Study IDs: 02-05-2025
Record Dates: First submitted 2025-07-11; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: the Detection of Prostate Cancer in Men

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PSA — Prostate-Specific Antigen test, a blood test used to measure the level of PSA in a man's blood. PSA is a protein produced by the prostate gland, and elevated levels can indicate various conditions, including prostate cancer, benign prostatic hyperplasia (BPH), or prostatitis.
Diagnostic Test: DRE — A digital rectal exam (DRE) is a procedure where a doctor inserts a lubricated, gloved finger into the rectum to check for abnormalities.

SUMMARY:
Prostate cancer is a significant health concern in the Middle East, including Syria, where many cases are diagnosed at advanced stages due to low awareness and inadequate screening practices. The mortality-to-incidence ratio for prostate cancer in the region is alarmingly high, indicating a pressing need for effective early detection strategies.

DETAILED DESCRIPTION:
This study aims to assess the awareness, attitudes, and practices regarding prostate cancer screening among men in the middle region of Syria, with the goal of identifying barriers to early detection and informing public health interventions.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 40 years and older residing in the middle region of Syria.

Exclusion Criteria:

* Men with a previous diagnosis of prostate cancer.

Ages: 40 Years to 65 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Detection of Prostate cancer in syrian men aged 40-65
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-05-17 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of ptients with early signs of prostate cancer | From Participant enrolment to the end of the study at 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Hawash Private University, Homs, Syria

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT07075666/Prot_SAP_000.pdf